CLINICAL TRIAL: NCT05206981
Title: IlluminOss Device Global Registry - A Prospective, Post-Market, Multi-Center Evaluation of the Clinical Outcomes of the IlluminOss Device
Brief Title: Device Global Registry for the IlluminOss Bone Stabilization System
Status: Recruiting | Type: Observational
Sponsor: IlluminOss Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REP-2012
Record Dates: First submitted 2022-01-08; First posted 2022-01-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Fracture; Pathological Fracture
MeSH Terms: conditions — Fractures, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: IlluminOss Device — Patients may enroll in the registry if they have been implanted (retrospective) or will be implanted (prospective) with the IlluminOss device.

SUMMARY:
This is a multi-center, observational patient registry. The primary objective of the study is to collect safety and performance data on the IlluminOss Device when used to provide stabilization and alignment for the treatment of traumatic or impending and pathologic fractures.

DETAILED DESCRIPTION:
This is a registry database which will collect patient data as part of a physician's standard of care. Medical data will be collected on patients via questionnaires in either web based or paper forms. Both prospective and retrospective data will be entered into the database. Data collection will begin during the initial visit to the clinic. Demographic, surgical, hospital discharge, and adverse event data will be collected as well as patient reported outcomes including the PROMIS physical function, Visual Analog Pain Score (VAS), and Veterans Rand 12 (VR 12) surveys. Patients will be asked to complete these surveys at the pre-operative and post operative visits at 75 days, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been deemed a candidate for the IlluminOss device
2. Patient is male or non-pregnant female
3. Patient is willing and able to comply with the postoperative scheduled clinical and radiographic evaluations
4. Patient is willing and able to give informed consent if required
5. Traumatic patient is over the age of 50
6. IlluminOss procedure is the initial procedure to treat the traumatic injury

Exclusion Criteria:

United States (U.S.)

This product is contraindicated in U.S. patients who have:

1. an active or incompletely treated infection that could involve the site where the device will be implanted;
2. are allergic to any of the implant materials or to dental glue;
3. have an intramedullary canal measuring smaller than the diameter of the delivery sheath provided at the site of the fracture;
4. distant foci of infections which may spread to the implant site, have open fractures with severe contamination;
5. or in patients for whom delivery sheath is unable to cross fracture site after proper fracture reduction and realignment.

European Union (EU)

This product is contraindicated in EU patients who have:

For all Bones:

1. Patients who are considered skeletally immature.
2. Presence of active or incompletely treated infections that could involve the site where the device will be implanted.
3. Patients allergic to any of the implant materials, or to dental glue.
4. Patients whose intramedullary canal at site of fracture measures smaller than the diameter of the sheath provided.
5. Uncooperative patient or patient with neurologic disorder, incapable of following directions.
6. Distant foci of infections which may spread to the implant site.
7. Vascular insufficiency.
8. Open fractures with severe contamination.
9. Extremely comminuted fractures where insufficient holding power of the balloon on the intramedullary canal is probable.
10. Delivery sheath is unable to cross fracture site after proper fracture reduction and realignment.

    For acute Humerus fractures:
11. Patients who are under the age of Fifty (50)

    For all bones excluding pathologic Humerus:
12. Metabolic disorders which may impair bone formation.
13. Osteomalacia.
14. Vascular insufficiency, muscular atrophy, or neuro-muscular disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary objective of the study is to collect safety and performance data on the IlluminOss Device when used to provide stabilization and alignment for the treatment of traumatic or impending and pathologic fractures. The device will be used in a manner consistent with the treating physician's regular clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite Safety Success Rate | 12 Months

SECONDARY OUTCOMES:
Complications/Adverse Events | 12 Months
Successful Device Implantation | 12 Months
Fracture Healing | 12 Months
Disability & Return to Work Status | 12 Months
Discharge Status | 12 Months
Visual Analog Pain Score | 12 Months
Veterans Rand 12 Item Health Survey | 12 Months
Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function | 12 Months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (13):
  - Gulf Orthopedics, Mobile, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Presbyterian St Luke's Medical Ctr, Denver, Colorado
  - University of Miami Hospital, Miami, Florida
  - Weston Outpatient Surgical Center, Weston, Florida
  - Parkview Health, Fort Wayne, Indiana
  - Jacobi Medical Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Ortho Rhode Island, Wakefield, Rhode Island
  - Memorial Hermann Hospital, Katy, Texas
- Germany (3):
  - St Vinzenz Hospital, Cologne
  - Johannes Wesling Hospital Minden, Minden
  - Petrus Hospital, Wuppertal

IPD SHARING:
Plan to Share IPD: No